CLINICAL TRIAL: NCT00175058
Title: Acute Myocardial Infarction With HyperOxemic Therapy II
Brief Title: Acute Myocardial Infarction With HyperOxemic Therapy II (AMIHOT II)
Acronym: AMIHOT II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMIHOT II
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Myocardial Infarction
Keywords: Heart Attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control - Patients with acute anterior myocardial infarction revascularized by means of PCI with stenting within 6 hours of onset of symptoms, no experimental intervention
- 2 (Experimental): AO Therapy group - anterior acute myocardial infarction patients revascularized by means of PCI with stenting within 6 hours of symptom onset, receiving adjunctive infusion of hyperoxemic blood into target coronary artery for 90 minutes post-PCI.
  Interventions: Device: AO Therapy (aqueous oxygen)

INTERVENTIONS:
Device: AO Therapy (aqueous oxygen) — 90-min adjunctive reperfusion of hyperoxemic blood into target coronary artery, immediately following revascularization by means of PCI with stenting
  Other Names: AO Therapy; SSO2 Therapy
  Arms: 2

SUMMARY:
To determine whether or not HyperOxemic therapy rendered to patients (that meet the study inclusion criteria) with anterior acute myocardial infarction < 6 hours from symptom onset to reperfusion, results in a significant reduction in infarct size as measured by SPECT @ 14 days post event.

DETAILED DESCRIPTION:
The AMIHOT II clinical trial is designed as a focused study of a promising patient subset from the completed AMIHOT study. A brief synopsis of the AMIHOT experience is provided below, followed by a description of the AMIHOT II study.

The pivotal AMIHOT clinical study for the TherOx® Aqueous Oxygen (AO) System in treating post acute myocardial infarction (AMI) patients was approved by FDA on January 10, 2002 under IDE G980257/S011. The study objective was to determine whether the adjunctive administration of AO Therapy immediately after successful PCI in a group of patients presenting less than 24 hours from AMI symptom onset improves left ventricular function and reduces the area of infarction, with no increased incidence of 30-day Major Adverse Cardiac Events (MACE) when compared to a control group receiving only PCI standard-of-care treatment. 30-day MACE comprises the combined incidence of death, reinfarction, target vessel revascularization, and stroke.

Two hundred eighty-nine (289) patients were enrolled from January 16, 2002 through December 24, 2003, including 20 run-in subjects and 269 randomized patients. Three independent biomarkers (infarct size reduction, regional wall motion score improvement at three months, and reduction in ST segment elevation) were designated as co-primary endpoints to evaluate the effectiveness of AO Therapy. The study was designed to demonstrate superiority of the AO Therapy group as compared to controls for each of these endpoints, and to demonstrate non-inferiority of the AO Therapy group as compared to Control with respect to 30-day MACE. The study population was comprised of qualifying AMI patients treated with either PCI alone or with AO Therapy as an adjunct to successful PCI within 24 hours of symptom onset.

The observed 30-day MACE rates were comparable between the AO Therapy and Control groups. The AMIHOT trial results revealed positive trends for the overall study population in favor of the AO Therapy test group in each of the three co-primary endpoints. These favorable results did not demonstrate the required level of statistical significance to claim superiority. However, an examination of a pre-specified patient subset, anterior AMI subjects treated within six hours of symptom onset, showed promising results after analysis of the surrogate endpoint data, forming the basis for this IDE supplement that requests approval to conduct a new trial focused on this further defined patient population.

TherOx has designed a follow-up clinical trial focused on these anterior AMI subjects treated within six hours, utilizing a Bayesian statistical design that incorporates both the existing AMIHOT data, and the new proposed AMIHOT II study data, into a hierarchical model for combined analysis.

The key differences between the proposed AMIHOT II study and the previously conducted AMIHOT trial are:

* Focused target patient population - anterior AMI subjects revascularized within six hours of symptom onset. (AMIHOT included patients revascularized within 24 hours of symptom onset, irrespective of location of infarct.)
* Single effectiveness endpoint - infarct size reduction as measured by 14-day Tc-99m Sestamibi SPECT imaging. (AMIHOT included 3 co-primary endpoints)
* Non-inferiority comparison of 30-day MACE rates within a 6% safety delta (AMIHOT proposed an 8% delta.)
* Randomization scheme - AMIHOT II will be randomized on a 2.8:1 (AO Therapy Group: Control Group) basis, as compared to the (1:1) randomization used in AMIHOT.

The method of administration of AO Therapy and the basic design of the AO System and AO Cartridge have not changed since the approval was granted by FDA to conduct the AMIHOT trial. The IDE number for the AMIHOT II clinical proposal is consistent with AMIHOT (G980257).

ELIGIBILITY:
INCLUSION CRITERIA

Candidates for this study must meet ALL of the following criteria:

Pre-PCI:

1. Patient must be >= 18 years of age
2. AMI must be anterior
3. Patient is experiencing clinical symptoms consistent with anterior AMI of < 6 hour duration from time of symptom onset until admission to the emergency room
4. Complete medical history, history of AMI, previous coronary interventions, list of medications given within last 24 hours
5. 12-lead qualifying ECG criteria: Anterior infarction (ST-segment elevation > 1 mm in two or more contiguous leads between V1 and V4 or new left bundle branch block (LBBB) with documentation of LAD system culprit lesion)
6. Patient provides written, Informed Consent
7. Patient and his/her physician agree to all required follow-up procedures and visits
8. Women of childbearing potential who have a negative pregnancy test (applies to female patients only)

   ANGIOGRAPHIC INCLUSION CRITERIA: These are evaluated after the subject has provided signed Informed Consent but prior to randomization:
9. Based on coronary anatomy, PCI is indicated for culprit lesion with anticipated use of an Intra-Coronary Stent
10. TIMI 0, I, or II flow is present on the initial angiographic injection of the infarct-related artery
11. Successful angioplasty as documented by < 50% diameter residual angiographic stenosis within and associated with the culprit lesion and ³ TIMI II flow and no major complications such as perforation or shock
12. Documented time of reperfusion is < 6 hours from the documented time of symptom onset

    EXCLUSION CRITERIA

    Candidates will be excluded from this study if ANY of the following conditions apply:

    Pre-PCI:
13. Patients with ventricular pseudoaneurysm, VSD, or papillary muscle rupture.
14. Absolute contraindications to anticoagulant therapy, including hemorrhagic diathesis or thrombocytopenia
15. Systemic Arterial pO2 is < 80 mmHg with supplemental oxygen
16. Placement of an intra-aortic balloon pump (IABP)
17. Patient has had coronary bypass surgery during the 30 day period preceding PCI
18. Severe known cardiac valvular stenosis or insufficiency, pericardial disease, or non-ischemic cardiomyopathy
19. Patients requiring cardiopulmonary resuscitation for > 10 minutes
20. Cardiogenic shock (SBP < 80 mm Hg for more than 30 minutes unresponsive to fluids or requiring intravenous pressors or placement of an IABP)
21. Expected survival of less than 6 months due to non-cardiac condition
22. Current participation in other investigational device or drug trials that have not finished the primary efficacy endpoint follow-up parameters
23. Patient has had a hemorrhagic stroke during the 6 month period preceding PCI
24. Physician discretion regarding unacceptability for enrollment

    ANGIOGRAPHIC EXCLUSION CRITERIA: These are evaluated after the subject has provided signed Informed Consent but prior to randomization:
25. Any proximal coronary diameter stenosis > 40 % that would restrict native flow with the Tracker-38 infusion catheter in place
26. Infarct-related vessels that are either saphenous vein grafts and/or small second order coronary vessels that do not supply significant areas of myocardium
27. Presence of a non-stented coronary dissection upon completion of the PCI procedure
28. Unprotected left main diameter stenosis > 60%
29. Severe target vessel calcification or tortuosity
30. Multi - vessel disease that in the judgment of the investigator is best treated with emergent or urgent CABG or additional PCI within 30 days
31. In the investigator's opinion, the target vessel is unsuitable for either placing the infusion catheter or treatment with PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
A single SPECT scan will be used to determine whether or not the treatment results in a significant reduction in infarct size in the treatment group. The scan is performed 14 days post-event. | 14 +/- 7 days
Safety will be determined by comparing 30-day MACE (Major Adverse Cardiac Events) rates, where MACE is comprised by the combined incidence of death, stroke, repeat MI, and target vessel revascularization. | 30 days

SECONDARY OUTCOMES:
ST elevation reduction will be compared between the two randomized groups at 3, 4, and 6 hours post-intervention | 3, 4, and 6 hrs post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Bryn Mawr Hospital, Bryn Mawr, Pennsylvania, United States

REFERENCES:
- [Derived] Stone GW, Martin JL, de Boer MJ, Margheri M, Bramucci E, Blankenship JC, Metzger DC, Gibbons RJ, Lindsay BS, Weiner BH, Lansky AJ, Krucoff MW, Fahy M, Boscardin WJ; AMIHOT-II Trial Investigators. Effect of supersaturated oxygen delivery on infarct size after percutaneous coronary intervention in acute myocardial infarction. Circ Cardiovasc Interv. 2009 Oct;2(5):366-75. doi: 10.1161/CIRCINTERVENTIONS.108.840066. Epub 2009 Sep 15. PMID 20031745